CLINICAL TRIAL: NCT00406003
Title: A Randomized, Open, Three-period Crossover Study to Compare the Pharmacokinetic Profile of Paroxetine After Single Dosing of Each Enteric-coated Geomatrix Control Release Tablet Strength (12.5, 25, 37.5mg) in Healthy Chinese Subjects
Brief Title: Single Dose Pharmacokinetic (PK) Study Of Paroxetine CR(12.5-37.5mg) In Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PCR104074
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Depressive Disorder
Keywords: BRL029060/Paroxetine CR; pharmacokinetics; safety
MeSH Terms: conditions — Depressive Disorder

ARMS (6):
- Subjects receiving treatment sequence ABC (Experimental): Eligible subjects will receive treatment sequence ABC; A= paroxetine 12.5 milligrams, B= paroxetine 25 milligrams, and C= paroxetine 37.5 milligrams separated by a wash-out period of 10 days.
  Interventions: Drug: Paroxetine controlled release tablet
- Subjects receiving treatment sequence BAC (Experimental): Eligible subjects will receive treatment sequence BAC; B= paroxetine 25 milligrams, A= paroxetine 12.5 milligrams and C= paroxetine 37.5 milligrams separated by a wash-out period of 10 days.
  Interventions: Drug: Paroxetine controlled release tablet
- Subjects receiving treatment sequence CBA (Experimental): Eligible subjects will receive treatment sequence CBA; C= paroxetine 37.5 milligrams, B= paroxetine 25 milligrams and A= paroxetine 12.5 milligrams separated by a wash-out period of 10 days.
  Interventions: Drug: Paroxetine controlled release tablet
- Subjects receiving treatment sequence BCA (Experimental): Eligible subjects will receive treatment sequence BCA; B= paroxetine 25 milligrams, C= paroxetine 37.5 milligrams and A= paroxetine 12.5 milligrams separated by a wash-out period of 10 days.
  Interventions: Drug: Paroxetine controlled release tablet
- Subjects receiving treatment sequence CAB (Experimental): Eligible subjects will receive treatment sequence CAB; C= paroxetine 37.5 milligrams, A= paroxetine 12.5 milligrams and B= paroxetine 25 milligrams separated by a wash-out period of 10 days.
  Interventions: Drug: Paroxetine controlled release tablet
- Subjects receiving treatment sequence ACB (Experimental): Eligible subjects will receive treatment sequence ACB; A= paroxetine 12.5 milligrams, C= paroxetine 37.5 milligrams and B= paroxetine 25 milligrams separated by a wash-out period of 10 days.
  Interventions: Drug: Paroxetine controlled release tablet

INTERVENTIONS:
Drug: Paroxetine controlled release tablet — Paroxetine will be given as single dose, controlled release tablet with dosing strengths of 12.5, 25 and 37.5 milligrams in fasted state separated by a wash-out period of 10 days.

SUMMARY:
The study was designed to describe the relationship between dose and pharmacokinetic parameters of paroxetine over the range of proposed dosage strengths of the paroxetine CR tablet (12.5 to 37.5 mg) as well as safety profile

ELIGIBILITY:
Inclusion criteria:

* 19-45 years healthy Chinese
* Body weight > 50 kg
* BMI between 19-25
* serological negative for HIV, syphilis and hepatitis B and C
* no abnormalities in ECG
* Female with negative pregnancy and male has no plan to have a child during and 3 months after the study.

Exclusion criteria:

* History of chronic physical/mental disease, current disease and concomitant medication

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2006-03-24 (Actual); Primary Completion 2006-04-26 (Actual); Study Completion 2006-04-26 (Actual)

PRIMARY OUTCOMES:
To obtain pharmacokinetic parameters of paroxetine paroxetine CR tablet (12.5 to 37.5 mg) in healthy Chinese subjects | Up to 32 days

SECONDARY OUTCOMES:
To describe Safety profile of healthy subjects when dosed with paroxetine controlled release | Up to 32 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Beijing, China

REFERENCES:
- See also: Results for study PCR104074 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/PCR104074?search=study&study_ids=PCR104074#rs